CLINICAL TRIAL: NCT06805396
Title: Timely Integration of Palliative Care in Oncology Care for Patients Referred for Palliative Radiotherapy on Bone Metastases: a Randomized Trial (TIPZO-RT Trial)
Brief Title: Timely Integration of Palliative Care in Oncology Care for Patients Referred for Palliative Radiotherapy on Bone Metastases: a Randomized Trial
Acronym: TIPZO-RT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roxanne Gal (Other)
Collaborators: Leiden University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Roxanne Gal, dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25U-0028
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Bone Metastases in Subjects with Advanced Cancer; Radiotherapy
Keywords: Palliative Care; Bone Metastases; Radiotherapy; Advanced Cancer; Quality of Life; Quality of Care

STUDY DESIGN:
Intervention Model Description: The trial will be conducted according to the Trials within Cohorts (TwiCs) design. Patients who provided broad consent to participate in the prospective PRESENT bone metastases cohort study, and who are eligible to participate in TIPZO-RT, will be randomized to either the intervention or control arm. Patients allocated to the intervention arm will be informed about the intervention and asked informed to undergo the intervention, which they can accept or refuse. Patients allocated to the control arm will not be informed, and their data from the cohort will be used comparatively.
Masking Description: Patients allocated to the control arm are not aware that they are part of this trial/the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palliative care consultation (Experimental): Timely referral to the palliative care consult team.
  Interventions: Behavioral: Palliative Care Consult
- Control (No Intervention): Patients will not be informed about the trial and will receive standard of care.

INTERVENTIONS:
Behavioral: Palliative Care Consult — Patients receive a regular consult (30-45 min) with the hospital palliative care consult team (PCCT) that is tailored to the preferences and needs of the individual patient. The following topics can be discussed: 1) physical symptoms, and, where appropriate, followed by recommendations for symptom management and transfer of handovers to the treating care team, 2) psychological, social and spiritual distress, followed by provision of counseling or referral to another specialist if needed, 3) goals of care to explore participants' values, preferences and needs (advance care planning), and 4) discussion about the needed follow-up of palliative care, and 5) care for caregivers. At baseline, patients receive a validated symptom questionnaire (Utrecht Symptom Diary (USD)-4D), which can be used as input for discussion during the consultation. If necessary, patients may have a follow up.
  Arms: Palliative care consultation

SUMMARY:
Rationale: With improvements in systemic tumour-directed treatments for primary tumours, survival rates for patients with bone metastases are improving. However, individual illness trajectories become less predictable and more vulnerable to adverse events from treatments, negatively impacting a patient's quality of life (QoL). Palliative care is aimed at reducing symptoms and improving QoL for patients with incurable diseases through early identification, thorough assessment, and effective management of physical, psychological, social, and spiritual challenges. Early integration of specialist palliative care into oncology care has shown to reduce symptom burden and potentially inappropriate end-of-life care, and to enhance QoL, yet it is often initiated late.

Objective: The primary objective is to evaluate the satisfaction with care and QoL experienced by patients with bone metastases who are offered a consultation with the hospital palliative care consultation team (PCCT) when referred for palliative radiotherapy compared to patients who receive standard of care.

Study design: A prospective, pragmatic, two-arm multicenter randomized controlled trial within the PRospective Evaluation of interventional StudiEs on boNe meTastases (PRESENT+) cohort that follows the Trials within Cohorts (TwiCs) design.

Study population: Patients with bone metastases referred for palliative radiotherapy who have their treating physician in one of the participating centers and have not been in contact with the hospital PCCT before.

Intervention: A consultation with the hospital PCCT within two weeks after inclusion in PRESENT+. In the standard of care control group, no consultation with the PCCT will be scheduled. They may have a consultation during follow-up if referring physicians may consider a consultation appropriate, or when patients themselves feel they want a referral.

Main study parameters/endpoints: Satisfaction with care (affective behavior) four weeks after inclusion in PRESENT+.

ELIGIBILITY:
Inclusion Criteria:

1. broad informed consent for PRESENT+ (i.e., consent for filling out questionnaires at regular intervals and randomization into future intervention studies), and
2. having their treating physician in the TIPZO-RT study site (UMC Utrecht, Radboudumc or LUMC).

Exclusion Criteria:

1. not able to understand the objective of the study (in Dutch),
2. cognitive impairment or dementia, and
3. has been in contact with palliative care consultants of the hospital PCCT before.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with care | 4 weeks after the start of radiotherapy
  Satisfaction with care is measured by the EORTC PATSAT-C33 - Affective behavior scale. The 33-item questionnaire includes three sections addressing the perceived quality of care provided by doctors, nurses/radiotherapy technicians, and service/care organization. Participants are asked to rate their experience for each item on a five-point Likert scale (poor to excellent). For this study, we use the 4-item affective behavior scale from the "nurses and radiotherapy technicians" section. Instead of rating "nurses and radiotherapy technicians", we ask the participants to rate the care from "healthcare providers" in the hospital to broadly assess patient satisfaction.

SECONDARY OUTCOMES:
Symptom burden | Baseline (start radiotherapy), after 4 and 8 weeks, and 3 and 6 months, and the BPI also after 2 and 6 weeks
  Symptom burden including physical, psychological, social and spiritual symptoms (Utrecht Symptom Diary (USD-)4D)
Pain | Baseline (start radiotherapy), after 4 and 8 weeks, and 3 and 6 months, and the BPI also after 2 and 6 weeks
  Pain as measured with the Brief Pain Inventory (BPI)
Quality of Life | Baseline (start radiotherapy), after 4 and 8 weeks, and 3 and 6 months
  QoL including physical and emotional functioning, and global QoL (EORTC QLQ-C15-PAL) and Painful Sites, Pain Characteristic, Functional Interference and Psychosocial Aspects (EORTC-QLQ-BM22)
Other satisfaction with care outcomes | Baseline (start radiotherapy), after 4 and 8 weeks, and 3 and 6 months
  Other satisfaction with care outcomes including information, coordination, and overall care (EORTC PATSAT-C33)
Overall survival | Max. two years
  Overall survival with a maximum follow-up of two years
Palliative care utilization | Through study completion, about 2 years
  Palliative care utilization: within the intervention group, we will measure the number of patients that were allocated to the intervention group and accepted referral (now or later in the disease trajectory) to the PCCT.
Palliative care utilization | Through study completion
  Palliative care utilization: within the intervention group, we will measure reasons for refraining from referral to the PCCT, e.g. too early, they think that they are not palliative, they expect no benefit, prior referral to the PCCT.
Palliative care utilization | Up to two years
  Palliative care utilization within the both the intervention and control group until death or up to two years post-randomization.

OTHER OUTCOMES:
Patient experiences and choices | Through study completion, about 2 years
  Semi-structured in-depth interviews with patients randomized to the intervention arm will be performed to obtain insight into patient experiences and choices regarding their consultations with the PCCT.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette M. van der Linden, Principal Investigator — Leiden University Medical Center; Natasja Raijmakers, Principal Investigator — Comprehensive Cancer Centre The Netherlands; Anouk van Oss, Principal Investigator — Leiden University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided